CLINICAL TRIAL: NCT01913262
Title: IFH Depression Registry 2013
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Institute for Family Health (Other)
Responsible Party: Principal Investigator, Virna Little, Senior Vice President of Psychosocial Services, The Institute for Family Health
Other Study IDs: IFH-DR-13
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Depression
Keywords: depression; phq9; phq-9; standard treatment
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months

GROUPS / COHORTS (1):
- IFH Patients on Depression Registry: Patients at the Institute for Family Health who have a diagnosis of depression active on their problem list or have had a diagnosis of depression used as an encounter diagnosis in the past year or patients with a PHQ-9 score greater than or equal to 10.
  Interventions: Behavioral: Standard Behavioral treatment

INTERVENTIONS:
Behavioral: Standard Behavioral treatment — Standard behavioral treatment (e.g. problem solving therapy, cognitive behavioral treatment)

SUMMARY:
This is an observational registry intended to track depression scores of patients over time in treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PHQ-9 score greater than or equal to 10, have a depression diagnosis active on the problem list, or have had a depression encounter diagnosis used in the past year, and are in behavioral health treatment at the Institute.

Exclusion Criteria:

* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community health patients in behavioral health treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Depression scores on PHQ-9 depression screening | 16 weeks
  Comparing depression scores for patients in treatment at initiation and after 16 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The Institute for Family Health, New York, New York, United States